CLINICAL TRIAL: NCT02550717
Title: A Pharmacoepidemiological Study on the Risk of Bleeding in New Users of Low-dose Aspirin (ASA) in The Health Improvement Network (THIN), UK
Brief Title: Epidemiological Study on the Safety of Aspirin in The Health Improvement Network (THIN)
Acronym: EPISAT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18116
Record Dates: First submitted 2015-09-03; First posted 2015-09-15 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Secondary Prevention; Stroke; Ischemic Heart Disease; Coronary Heart Disease
Keywords: Low-dose Acetylsalicylic Acid,; Bleeding,; The Health Improvement Network (THIN),; Cardiovascular; Secondary prevention of cardiovascular events
MeSH Terms: conditions — Stroke; Myocardial Ischemia; Coronary Disease; Hemorrhage | interventions — Aspirin; Clopidogrel; Anticoagulants; Anti-Inflammatory Agents, Non-Steroidal; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acetylsalicylic Acid: New users of low-dose Acetylsalicylic Acid (ASA)
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)
- Other medications: Users of other medications such as clopidogrel, oral anticoagulants, non-steroidal anti-inflammatory drugs (NSAIDs) and selective serotonin reuptake inhibitors (SSRIs)
  Interventions: Drug: Clopidogrel, Oral Anticoagulants, NSAIDs and SSRIs

INTERVENTIONS:
Drug: Acetylsalicylic Acid (Aspirin, BAYE4465) — Low-dose ASA for secondary prevention of cardiovascular events
  Groups: Acetylsalicylic Acid
Drug: Clopidogrel, Oral Anticoagulants, NSAIDs and SSRIs — Secondary prevention of cardiovascular events
  Groups: Other medications

SUMMARY:
To investigate the risk of major bleeding (including gastrointestinal and intracranial bleeding episodes) among new users of low-dose acetylsalicylic acid (ASA) in clinical practice

DETAILED DESCRIPTION:
These will be based on population-based cohorts using data from a primary care database in the UK: The Health Improvement Network (THIN) and will serve to make a clinically meaningful benefit-risk assessment regarding major bleeding consequences of ASA exposure in general population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-84 years
* Enrolled with the Primary Care Physician (PCP) for at least 2 years,
* To have a history of computerized prescriptions for at least 1 year prior
* To have at least one encounter/visit recorded in the last three years

Exclusion Criteria:

* To be exposed to low dose ASA before entering in the study
* Having a diagnosis of cancer before entering in the study
* Having a diagnosis of alcohol abuse before entering in the study
* Having a diagnosis of coagulopathies before entering in the study
* Having a diagnosis of esophageal varices before entering in the study
* Having a diagnosis of chronic liver disease before entering in the study

Ages: 40 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: THIN is a computerized medical research database that contains systematically recorded data on more than 3 million UK primary care patients. It is representative of this population with regard to age, sex, and geographic distribution, and has been validated for use in pharmacoepidemiological and epidemiological research in multiple studies 13. Participating Primary Care Physicians (PCPs) record prospectively data as part of their routine patient care, including demographics and life style factors (e.g. alcohol use, body mass index (BMI) and smoking status), consultation rates, referrals, hospital admissions, laboratory test results, diagnoses, prescriptions ordered by the PCPs, and a free text section, and send their data anonymously to THIN for use in research projects.
Sampling Method: Non-Probability Sample
Enrollment: 398158 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Intracranial bleeding among new users of low-dose Acetylsalicylic acid (ASA). | Up to 13 years
Incidence of Upper gastrointestinal bleeding among new users of low-dose ASA. | Up to 13 years
Incidence of Lower gastrointestinal bleeding among new users of low-dose ASA | Up to 13 years
Time to Intracranial bleeding among new users of low-dose ASA | Up to 13 years
Time to Upper gastrointestinal bleeding among new users of low-dose ASA | Up to 13 years
Time to Lower gastrointestinal bleeding among new users of low-dose ASA | Up to 13 years
Relative risk of Intracranial bleeding among new users of low dose ASA | Up to 13 years
  Relative risk is calculated as incident rate ratio produced by dividing the incidence rate of the outcome of interest in the exposed category by the incidence rate of the outcome of interest in the unexposed.
Relative risk of Upper gastrointestinal bleeding among new users of low-dose ASA | Up to 13 years
  Relative risk is calculated as incident rate ratio produced by dividing the incidence rate of the outcome of interest in the exposed category by the incidence rate of the outcome of interest in the unexposed.
Relative risk of Lower gastrointestinal bleeding among new users of low-dose ASA | Up to 13 years
  Relative risk is calculated as incident rate ratio produced by dividing the incidence rate of the outcome of interest in the exposed category by the incidence rate of the outcome of interest in the unexposed.

SECONDARY OUTCOMES:
Relative risk of Intracranial bleeding associated with use of other medications. | Up to 13 years
  Relative risk is calculated as incident rate ratio produced by dividing the incidence rate of the outcome of interest in the exposed category by the incidence rate of the outcome of interest in the unexposed.To estimate relative risk in users of other medications such as clopidogrel,oral anticoagulants, non-steroidal anti-inflammatory drugs (NSAIDs) and selective serotonin reuptake inhibitors (SSRIs), independently from use of low-dose ASA and concomitantly
Relative risk of Upper gastrointestinal bleeding associated with use of other medications | Up to 13 years
  Relative risk is calculated as incident rate ratio produced by dividing the incidence rate of the outcome of interest in the exposed category by the incidence rate of the outcome of interest in the unexposed.To estimate relative risk in users of other medications such as clopidogrel,oral anticoagulants, non-steroidal anti-inflammatory drugs (NSAIDs) and selective serotonin reuptake inhibitors (SSRIs), independently from use of low-dose ASA and concomitantly
Relative risk of Lower gastrointestinal bleeding associated with use of other medications. | Up to 13 years
  Relative risk is calculated as incident rate ratio produced by dividing the incidence rate of the outcome of interest in the exposed category by the incidence rate of the outcome of interest in the unexposed.To estimate relative risk in users of other medications such as clopidogrel,oral anticoagulants, non-steroidal anti-inflammatory drugs (NSAIDs) and selective serotonin reuptake inhibitors (SSRIs), independently from use of low-dose ASA and concomitantly

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, United Kingdom

REFERENCES:
- [Result] Cea Soriano L, Gaist D, Soriano-Gabarro M, Bromley S, Garcia Rodriguez LA. Low-dose aspirin and risk of intracranial bleeds: An observational study in UK general practice. Neurology. 2017 Nov 28;89(22):2280-2287. doi: 10.1212/WNL.0000000000004694. Epub 2017 Nov 1. PMID 29093065
- [Result] Cea Soriano L, Gaist D, Soriano-Gabarro M, Garcia Rodriguez LA. Incidence of intracranial bleeds in new users of low-dose aspirin: a cohort study using The Health Improvement Network. J Thromb Haemost. 2017 Jun;15(6):1055-1064. doi: 10.1111/jth.13686. Epub 2017 May 2. PMID 28371181